CLINICAL TRIAL: NCT03085043
Title: Magnetic Resonance Imaging as a Comprehensive Staging Tool for the Evaluation of High-Risk Prostate Carcinoma
Brief Title: Magnetic Resonance Whole Body Diffusion-Weighted Imaging in Finding Bone or Lymph Node Metastasis in Participants With High-Risk Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2015-0053; NCI-2018-01308 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0053 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2017-03-15; First posted 2017-03-21 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (bone scan, CT, MRI, magnetic resonance WB-DWI) (Experimental): Participants undergo standard of care bone scan, CT of the abdomen and pelvis, and pelvic MRI. Participants also undergo magnetic resonance WB-DWI over 20-30 minutes.
  Interventions: Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Magnetic Resonance Whole Body Diffusion-Weighted Imaging

INTERVENTIONS:
Procedure: Bone Scan — Undergo bone scan
Procedure: Computed Tomography — Undergo CT of the abdomen and pelvis
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Procedure: Magnetic Resonance Imaging — Undergo pelvic MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Magnetic Resonance Whole Body Diffusion-Weighted Imaging — Undergo magnetic resonance whole body diffusion-weighted imaging
  Other Names: WB DW MRI; WB-DWI; Whole Body Magnetic Resonance Imaging Using Diffusion-Weighted Images; Whole-Body Diffusion-Weighted MRI

SUMMARY:
This trial studies how well magnetic resonance whole body diffusion-weighted imaging works in finding cancer that has spread to the bone or lymph nodes (metastasis) in participants with high-risk prostate cancer. Diagnostic procedures, such as magnetic resonance whole body diffusion-weighted imaging (a method to show how water moves in a certain area) may help find bone or lymph nodes metastasis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare accuracies of whole body magnetic resonance imaging (MRI) versus bone scan plus computed tomography (CT) scan in detecting bone or lymph node metastasis in high risk prostate cancer patients.

OUTLINE:

Participants undergo standard of care bone scan, CT of the abdomen and pelvis, and pelvic MRI. Participants also undergo magnetic resonance whole body (WB)-diffusion-weighted imaging (DWI) over 20-30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Prostate carcinoma patients at high risk for metastasis with prostate-specific antigen (PSA) more than 20 ng/ml and/or Gleason score = 8/ > 8.
* Ability to understand and sign informed consent.

Exclusion Criteria:

* Patient is at low risk for metastasis with Gleason score at diagnosis < 8.
* Currently receiving or history of systemic therapy with testosterone suppressing medication (i.e., lupron, degarelix, abiraterone, enzalutamide) or local radiation therapy.
* Contraindication to magnetic resonance imaging (MRI).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2016-04-20 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of whole body magnetic resonance imaging (MRI) | Up to 6 months
  Accuracy will be estimated along with 95% confidence intervals for whole body MRI (for bone and lymph node metastasis), bone scan (for bone metastasis), and computed tomography (CT) scan (for lymph node metastasis). Comparisons between modalities will be performed using McNemar's test. Other statistical analyses will be carried out as appropriate.

SECONDARY OUTCOMES:
Sensitivity of MRI, bone scan, and CT scan | Up to 9 years
  Sensitivity will be estimated along with 95% confidence intervals for whole body MRI (for bone and lymph node metastasis), bone scan (for bone metastasis), and CT scan (for lymph node metastasis). Comparisons between modalities will be performed using McNemar's test. Other statistical analyses will be carried out as appropriate.
Specificity of MRI, bone scan, and CT scan | Up to 9 years
  Specificity will be estimated along with 95% confidence intervals for whole body MRI (for bone and lymph node metastasis), bone scan (for bone metastasis), and CT scan (for lymph node metastasis). Comparisons between modalities will be performed using McNemar's test. Other statistical analyses will be carried out as appropriate.
Positive predictive value (PPV) of MRI, bone scan, and CT scan | Up to 9 years
  PPV will be estimated along with 95% confidence intervals for whole body MRI (for bone and lymph node metastasis), bone scan (for bone metastasis), and CT scan (for lymph node metastasis). Comparisons between modalities will be performed using McNemar's test. Other statistical analyses will be carried out as appropriate.
Negative predictive value (NPV) of MRI, bone scan, and CT scan | Up to 9 years
  NPV will be estimated along with 95% confidence intervals for whole body MRI (for bone and lymph node metastasis), bone scan (for bone metastasis), and CT scan (for lymph node metastasis). Comparisons between modalities will be performed using McNemar's test. Other statistical analyses will be carried out as appropriate.
Detection of other types of metastases | Up to 9 years
  Comparisons between modalities will be performed using McNemar's test. Other statistical analyses will be carried out as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Tharakeswara K Bathala, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org